CLINICAL TRIAL: NCT00815269
Title: Vasodilation Effect of Inhalational Anesthetics Including Halothane, Isoflurane, Sevoflurane, Desflurane and Enflurane
Brief Title: Vasodilation Effect of Inhalational Anesthetics
Acronym: VEFIHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMU-200812-MZ39; NJFY0812015
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: General Anesthesia
Keywords: Inhalant anesthetic; Vasodilation; General anesthesia; Ultrasonography
MeSH Terms: conditions — Aneurysm | interventions — Halothane; Isoflurane; Sevoflurane; Desflurane; Enflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Active Comparator): Halothane anesthesia: induction and maintenance with different doses
  Interventions: Drug: Halothane
- 2 (Experimental): Isoflurane anesthesia: induction and maintenance with different doses
  Interventions: Drug: Isoflurane
- 3 (Experimental): Sevoflurane anesthesia: induction and maintenance with different doses
  Interventions: Drug: Sevoflurane
- 4 (Experimental): Desflurane anesthesia: induction and maintenance with different doses
  Interventions: Drug: Desflurane
- 5 (Experimental): Enflurane anesthesia: induction and maintenance with different doses
  Interventions: Drug: Enflurane

INTERVENTIONS:
Drug: Halothane — Induction: 2-4% halothane pluses 3-5 L/min oxygen Maintenance: different doses from 0.5% to 3% with 1-2 L/min oxygen
  Other Names: Fluothane
  Arms: 1
Drug: Isoflurane — Induction: 2-5% isoflurane pluses 3-5 L/min oxygen Maintenance: different doses from 1% to 4% with 1-2 L/min oxygen
  Other Names: Forane
  Arms: 2
Drug: Sevoflurane — Induction: 3-8% sevoflurane pluses 3-5 L/min oxygen Maintenance: different doses from 1% to 4% with 1-2 L/min oxygen
  Other Names: Sevorane
  Arms: 3
Drug: Desflurane — Induction: 2-8% desflurane pluses 3-5 L/min oxygen Maintenance: different doses from 1% to 4% with 1-2 L/min oxygen
  Other Names: Suprane
  Arms: 4
Drug: Enflurane — Induction: 2-5% enflurane pluses 3-5 L/min oxygen Maintenance: different doses from 1% to 4% with 1-2 L/min oxygen
  Other Names: Ethrane
  Arms: 5

SUMMARY:
Previous studies on animals suggest that inhalational anesthetics can reduce vascular tension in vitro resulting in vasodilation and decrease in blood pressure. This role for inhalational anesthetics has essential clinical implications such as the condition of sepsis or septic shock or other shock-associated states during which the blood vessel constricts strongly and leads to circulation dysfunction. The vasodilation property of these anesthetics including halothane, isoflurane, sevoflurane, desflurane and enflurane enables them to be better options than other general anesthetics in many clinical conditions needing the vasculature to be dilated. The investigators hypothesized that these inhalational anesthetics can evoke vasodilation measured with ultrasonography during general anesthesia in vivo as the in vitro studies displayed.

ELIGIBILITY:
Inclusion Criteria:

* Must be undergoing general anesthesia
* Age between 19-45 years

Exclusion Criteria:

* With hypertension
* Existing organic dysfunction
* Allergic to inhalant anesthetics
* Alcohol addictive or narcotic dependent patients
* A history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Ultrasonography of blood vessels including radial artery, brachial artery, femoral artery, popliteal artery | Ten min prior to anesthesia; 0 min of anesthesia; 0 min of the end of anesthesia induction; 5, 10, 20, 30, 60 min during maintenance of the anesthesia

SECONDARY OUTCOMES:
Blood flow volume during anesthesia of the vasculature | Ten min prior to anesthesia; 0 min of anesthesia; 0 min of the end of anesthesia induction; 5, 10, 20, 30, 60 min during maintenance of the anesthesia
Blood pressure including systolic, diastolic and mean artery blood pressures | Ten min prior to anesthesia; 0 min of anesthesia; 0 min of the end of anesthesia induction; 5, 10, 20, 30, 60 min during maintenance of the anesthesia
The time interval of between the initiation of the inhalational anesthetics delivered to the beginning of decreasing of blood pressure | From the beginning of anesthesia (0 min) till the first time of blood pressure decreased, this measure would be varied according to different individuals
The total dose of phenylephrine required to maintain baseline arterial blood pressure | From the beginning of anesthesia (0 min) to 20 min after anesthesia begun
Regression and correlation analyses between different doses of the anesthetics and the extent of vasodilation | Forty eight hours after operation

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China